CLINICAL TRIAL: NCT01871532
Title: A Multi-Centre, Two-Arm, Interventional, Phase IV Study to Evaluate Tailoring of Recombinant FSH Treatment in Subjects With Chronic Anovulation Using the Gonal-f® Prefilled Pen in Women Undergoing Ovulation Induction
Brief Title: Low-dose Gonal-f® in Ovulation Induction
Acronym: LoGo
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was terminated because of delays in sourcing replacement Investigational Medicinal Product for the study due to manufacturing delays.
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR700623_535; 2012-003227-38 (EudraCT Number)
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Results first posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-06

CONDITIONS: Infertility; Monofollicular Development
Keywords: Monofollicular Development; Gonal-f®; Recombinant Follicle Stimulating Hormone; Ovarian hyperstimulation syndrome (OHSS)
MeSH Terms: conditions — Infertility; Ovarian Hyperstimulation Syndrome | interventions — follitropin alfa; Glycoprotein Hormones, alpha Subunit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Dose Gonal-f® Protocol (Experimental): Gonal-f was administered subcutaneously daily at a starting dose of 50 International unit (IU) for Week 1, then dose was gradually increased by 12.5 IU for two weeks, with a final increase of 25 IU, up to maximum dose of 100 IU, until Week 4 for subjects with minimal response. After adequate follicular development was achieved, the subject was administration human chorionic gonadotropin (hCG) within 24-48 hours of last Gonal-f injection as per investigator discretion.
  Interventions: Drug: Gonal-f®
- Standard Low Dose Gonal-f® Protocol (Active Comparator): Gonal-f was administered subcutaneously daily at a starting dose of 50 International Units (IU) for Week 1, then dose was gradually increased by 12.5 IU for two weeks, up to maximum dose of 125 IU, until Week 4 for subjects with minimal response. After adequate follicular development was achieved, the subject was administration human chorionic gonadotropin (hCG) within 24-48 hours of last Gonal-f injection as per investigator discretion.
  Interventions: Drug: Gonal-f®

INTERVENTIONS:
Drug: Gonal-f®
  Other Names: Recombinant follicle stimulating hormone (r-FSH)

SUMMARY:
This is a prospective, multicenter, open-label, comparative and parallel-group study of ovulation induction evaluating tailoring of Recombinant follicle stimulating hormone (FSH) treatment using the Gonal-f® prefilled pen in World Health Organization (WHO) Type 2 anovulatory subjects who have previously failed to conceive with clomifene treatment.

DETAILED DESCRIPTION:
Subjects will enter a screening period of up to one month before being randomized at the Baseline Visit, which will occur on Day 1 of the subject's menstrual cycle. Each subject will then receive up to 4 weeks treatment with Gonal-f®. If adequate follicular development (assessed by transvaginal ultrasound) is achieved, the subject will proceed to administration of human chorionic gonadotropin (hCG) within 24-48hrs of last Gonal-f® injection (or according to standard site practice).

Following administration of hCG, subjects will attempt to become pregnant via intercourse or intrauterine insemination. The method of conception will be determined by the subject's requirements and standard practice at the clinic site.

All subjects will be followed up appropriately until confirmation of biochemical pregnancy (hCG + minimum 14 days) and clinical pregnancy (hCG + minimum 42 days, for subjects with positive biochemical pregnancy test).

ELIGIBILITY:
Inclusion Criteria:

* Subjects eligible for ovulation induction treatment, where monofollicular development is the desired treatment outcome and the dose schedule outlined in the protocol is deemed appropriate
* Premenopausal female subjects, aged between 18 and 37 years inclusive
* Subjects desirous of pregnancy/willing to conceive
* Subjects who are infertile due to chronic anovulation demonstrated by cycle duration of greater than 35 days.
* Subjects who have been treated with clomifene citrate therapy, according to standard site practice, and have failed to ovulate and/or conceive
* Subjects with follicle stimulating hormone (FSH) and prolactin (PRL) serum values within the normal range in the early follicular phase
* Subjects with an overall total antral follicle count greater than 10 (of follicle size greater than or equal to 2 millimeter [mm] and less than 11 mm) (that is, total between both ovaries)
* Subjects with at least one patent tube, as documented by recent (within 2 years before treatment assignment) hysterosalpingography (HSG) or hysterosalpingo contrast sonography (HyCoSy)
* Subjects with normal uterine cavity, as documented by recent (within 2 years before treatment assignment) hysteroscopy, HSG or ultrasound scan
* Subjects with body mass index (BMI) greater than 20 and less than or equal to 32 kilogram per square meter (kg/m^2) (BMI is equal to body weight [kilogram {kg}] divided by Height * Height [square meter {m^2}])
* Subjects with negative cervical Papanicolaou (PAP) test conducted according to national guidelines and/or standard site practice
* Male partners of female subjects with sperm compatible with non-assisted fertilization or availability of donor sperm, as confirmed by the Investigator
* Subjects who are willing and able to comply with protocol requirements and have provided written, informed consent

Exclusion Criteria:

* Subjects with history of hypersensitivity to the investigational medicinal product (IMP) (active substance follitropin alpha, FSH, or to any of the excipients of Gonal-f®) or any other drug used in the trial (that is, Ovitrelle)
* Subjects with ovarian enlargement or ovarian cyst unrelated to Polycystic Ovary Syndrome (PCOS), and of unknown origin on ultrasound
* Subjects with evidence of diminished ovarian reserve (cycle length less than 26 days; FSH above the upper limit of local serum FSH values, total antral follicle count [AFC] in both ovaries less than 10)
* Subjects with uterine pathology/abnormalities, which in the opinion of the Investigator could impair pregnancy evolution
* Subjects who have undergone three or more previous miscarriages
* Subjects with any previous extrauterine pregnancy
* Pregnant or lactating female subjects
* Subjects with abnormal gynecological bleeding of unknown etiology.
* Subjects with previous history of severe ovarian hyper stimulation syndrome (OHSS) (after clomifene treatment)
* Subjects who have evidence of current or previous pelvic inflammatory disease before treatment assignment
* Subjects with tumors of the hypothalamus and pituitary gland
* Subjects with ovarian, uterine or mammary carcinoma
* Subjects treated with clomifene citrate or gonadotropins within 1 month of the screening evaluation
* Subjects with any medical condition which, in the opinion of the Investigator, would prevent an effective response, such as primary ovarian failure, or malformations of the reproductive organs incompatible with pregnancy
* Subjects with any medical condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the drug
* Subjects with any clinically significant systemic disease (for example, insulin-dependent diabetes) or any contraindication to being pregnant and/or carrying a pregnancy to term
* An active substance abuser
* Known infection with human immunodeficiency virus (HIV), Hepatitis B or C virus in the trial subject or her male partner
* Subjects who are currently participating in another clinical trial
* Subjects who are unable to give written informed consent

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono Limited, UK
Locations (10):
- Ireland (3):
  - Research Site, Cork
  - Research Site, Dublin
  - Research Site, Galway
- United Kingdom (7):
  - Research Site, Cambridge
  - Research site, Cheshunt
  - Research Site, Derby
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research site, London
  - Research Site, Nottingham

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose Gonal-f: Gonal-f was administered subcutaneously daily at a starting dose of 50 International unit (IU) for Week 1, then dose was gradually increased by 12.5 IU for two weeks, with a final increase of 25 IU, up to maximum dose of 100 IU, until Week 4 for subjects with minimal response. After adequate follicular development was achieved, the subject was administration human chorionic gonadotropin (hCG) within 24-48 hours of last Gonal-f injection as per investigator discretion.
- Standard Low Dose Gonal-f: Gonal-f was administered subcutaneously daily at a starting dose of 50 International Units (IU) for Week 1, then dose was gradually increased by 12.5 IU for two weeks, up to maximum dose of 125 IU, until Week 4 for subjects with minimal response. After adequate follicular development was achieved, the subject was administration human chorionic gonadotropin (hCG) within 24-48 hours of last Gonal-f injection as per investigator discretion.
Period: Overall Study
Arm/Group | Low Dose Gonal-f | Standard Low Dose Gonal-f
Started | 12 | 12
Subjects Received hCG Treatment | 11 | 9
Completed | 11 | 10
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) included all subjects randomized and that had received at least 1 Gonal-f injection and had number of follicles measured at any point.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Gonal-f | Standard Low Dose Gonal-f | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (2.96) | 29.5 (3.75) | 30.1 (3.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Cycles With Monofollicular Development
Description: The monofollicular development was defined as the number of cycles with monofollicular development only one Follicle Greater Than or Equal (>= to 17 millimeter (mm) and no other follicles Greater than or equal to 14 mm following up to 4 weeks Gonal-f treatment.
Time Frame: Baseline up to 4 weeks
Population: Data was not assessed since the study was terminated early due to the delay in providing additional study drug following a batch recall.
Arm/Group | Low Dose Gonal-f | Standard Low Dose Gonal-f
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Cycles With Bifollicular Development
Description: The bifollicular development was defined as the number of cycles with bifollicular development of only two follicles greater than or equal to 17 millimeter.
Time Frame: Baseline up to 4 weeks
Population: as for outcome 1
Arm/Group | Low Dose Gonal-f | Standard Low Dose Gonal-f
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Cycles With Multifollicular Development
Description: The multifollicular development was defined as the number of cycles with multifollicular development of three or more follicles greater than or equal to 14 millimeter
Time Frame: Baseline up to 4 weeks
Population: as for outcome 1
Arm/Group | Low Dose Gonal-f | Standard Low Dose Gonal-f
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Ovulatory Cycles
Description: Ovulation was defined as a serum progesterone (P4 ) level greater than or equal to 10 nanogram per milliliter (ng/mL) or Clinical Pregnancy. Clinical pregnancy was defined as pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy. It excludes ectopic pregnancy.
Time Frame: Baseline up to 42 days post human chorionic gonadotrophin (hCG) administration
Population: as for outcome 1
Arm/Group | Low Dose Gonal-f | Standard Low Dose Gonal-f
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Cycles Wherein Human Chorionic Gonadotropin (hCG) Was Not Administered
Time Frame: Baseline up to 4 weeks
Population: as for outcome 1
Arm/Group | Low Dose Gonal-f | Standard Low Dose Gonal-f
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Cycles Resulting in Clinical Pregnancy
Description: Clinical pregnancy was defined as pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy. It excludes ectopic pregnancy.
Time Frame: 35-42 days post hCG administration
Population: as for outcome 1
Arm/Group | Low Dose Gonal-f | Standard Low Dose Gonal-f
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Multiple Pregnancy
Description: Multiple pregnancy is a pregnancy where more than one fetus develops simultaneously in the womb. There are two types of twinning-identical and fraternal. Identical twins represent the splitting of a single fertilized zygote (union of two gametes or male/female sex cells that produce a developing fetus) into two separate individuals.
Time Frame: 35-42 days post hCG administration
Population: as for outcome 1
Arm/Group | Low Dose Gonal-f | Standard Low Dose Gonal-f
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Fetuses
Time Frame: 35-42 days post hCG administration
Population: as for outcome 1
Arm/Group | Low Dose Gonal-f | Standard Low Dose Gonal-f
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Miscarriages After Confirmation of Clinical Pregnancy
Description: Miscarriages were calculated per clinical pregnancy, and clinical pregnancy was defined as pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or confirmed by clinical signs of pregnancy. It excludes ectopic pregnancy.
Time Frame: 35-42 days post hCG administration
Population: as for outcome 1
Arm/Group | Low Dose Gonal-f | Standard Low Dose Gonal-f
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Subjects With Ovarian Hyper Stimulation Syndrome (OHSS)
Description: OHSS was defined as an exaggerated systemic response to ovarian stimulation characterized by a wide spectrum of clinical and laboratory manifestations, classified as mild, moderate or severe according to the degree of abdominal distention, ovarian enlargement and respiratory, hemodynamic and metabolic complications.
Time Frame: up to 42 days post hCG administration
Population: Safety population included all subjects who were randomised and received at least 1 Gonal-f injection.
Measure: Number; unit: subjects
Arm/Group | Low Dose Gonal-f | Standard Low Dose Gonal-f
Number analyzed (Participants) | 12 | 12
subjects | 0 | 0

11. Secondary Outcome: Duration of Recombinant Follicle Stimulating Hormone (rFSH) Stimulation
Time Frame: Baseline up to 4 weeks
Population: as for outcome 1
Arm/Group | Low Dose Gonal-f | Standard Low Dose Gonal-f
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Total Dose of Recombinant Follicle Stimulating Hormone (r-FSH) Administered Per Cycle
Time Frame: Baseline up to 4 weeks
Population: as for outcome 1
Arm/Group | Low Dose Gonal-f | Standard Low Dose Gonal-f
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline in Anti-Mullerian Hormone (AMH) Levels at Week 4
Time Frame: Baseline, Week 4
Population: as for outcome 1
Arm/Group | Low Dose Gonal-f | Standard Low Dose Gonal-f
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Testosterone Levels
Time Frame: Baseline
Population: as for outcome 1
Arm/Group | Low Dose Gonal-f | Standard Low Dose Gonal-f
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Sex Hormone Binding Globulin (SHBG) Levels
Time Frame: Baseline
Population: as for outcome 1
Arm/Group | Low Dose Gonal-f | Standard Low Dose Gonal-f
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Low Dose Gonal-f | Standard Low Dose Gonal-f
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/12
Other Adverse Events (participants affected / at risk) | 2/12 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Gonal-f (N=12) | Standard Low Dose Gonal-f (N=12)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Gonal-f (N=12) | Standard Low Dose Gonal-f (N=12)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Study was terminated because of delays in sourcing replacement Investigational Medicinal Product (IMP) for the study due to manufacturing delays hence the outcome measure was not assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other